CLINICAL TRIAL: NCT00002551
Title: Postoperative Evaluation of 5-FU by Bolus Injection vs. 5-FU by Prolonged Venous Infusion Prior to and Following Combined Prolonged Venous Infusion Plus Pelvic XRT vs. Bolus 5-FU Plus Leucovorin Plus Levamisole Prior to and Following Combined Pelvic XRT Plus Bolus 5-FU Plus Leucovorin in Patients With Rectal Cancer, Phase III
Brief Title: SWOG-9304 Chemotherapy Plus Radiation Therapy in Treating Patients With Rectal Cancer That Has Been Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Radiation Therapy Oncology Group (Network); North Central Cancer Treatment Group (Network); NCIC Clinical Trials Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000063349; SWOG-9304 (Other: SWOG); CAN-NCIC-CO11 (Other: NCIC); NCCTG-934751 (Other: NCCTG); RTOG-9403 (Other: RTOG); CLB-C9491 (Other: CALGB); INT-0144 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Levamisole; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bolus 5-FU, Pelvic XRT + PVI 5-FU, Bolus 5-FU (Experimental): Bolus 5-FU (fluorouracil) (500mg/m2/day on days 1-5, 29-33), Pelvic XRT + PVI 5-FU, Bolus 5-FU (450mg/m2/day for 5 days beginning 28 days after RT, for 2 cycles on days 1-5 of a 28 days cycle).
  Interventions: Drug: fluorouracil; Radiation: radiation therapy
- PVI 5-FU+Pelvic XRT+PVI 5-FU+PVI 5-FU (Experimental): 5-FU (fluorouracil) 300mg/m2/day for 42 days followed by 2 week interruption, Day 57 through XRT will receive 225mg/m2/day of 5-FU followed by 1 month interruption, 4 weeks after completion of XRT 1 8wk cycle of 5-FU 300mg/m2/day.
  Interventions: Drug: fluorouracil; Radiation: radiation therapy
- Bol 5-FU+LV+LEV+Pel XRT+Bol 5-FU+LV Bol 5-FU + LV + LEV (Experimental): 5-FU (fluorouracil) 425/mg/m2/day Days 1-5,29-33; LV (leucovorin calcium) 20mg/m2/day Days 1-5,29-33; LEV (levamisole hydrochloride) 150mg/day (50mg TID) for 3 days every 14 days starting after each course of 5-FU. During RT: 5-FU and LV 4 days on wk 1 and wk 5 of RT. LV 20 mg/m2/day IV bolus within 2hrs after completion of that day's radiation therapy, for four days in each cycle. Followed immediately by 5- FU 400 mg/m2/day IV bolus. Treatment will be given on days 57 - 60 and 85 - 88.Treatment post-RT-chemotherapy 28 days after completion of RT consist of 5 days of chemotherapy in 28 day cycles. 5-FU, 380 mg/m2/day on days 1 - 5 and LV given at a dose of 20 mg/m2/day on days 1 - 5 with the 5-FU given immediately after the LV. For 2 post-radiation cycles on days 1 - 5 of a 28 day cycle. Levamisole will be given orally at a dose of 150 mg/day (50 mg tid) for 3 days every 14 days during the 1st 3 days of each cycle of 5-FU, and again 14 days after starting each course of 5-FU.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: levamisole hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil — See arm assignments.
  Other Names: 5-FU
Drug: leucovorin calcium — See arm assignments.
  Other Names: leucovorin; LV
  Arms: Bol 5-FU+LV+LEV+Pel XRT+Bol 5-FU+LV Bol 5-FU + LV + LEV
Drug: levamisole hydrochloride — See arm assignments.
  Other Names: LEV
  Arms: Bol 5-FU+LV+LEV+Pel XRT+Bol 5-FU+LV Bol 5-FU + LV + LEV
Radiation: radiation therapy — See arm assignments.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which treatment regimen is more effective for rectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of combination chemotherapy plus radiation therapy in treating patients who have rectal cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall and relapse free survival of patients with stage II or III rectal cancer treated with one of the following three regimens: bolus injections of fluorouracil (5-FU) prior to and following pelvic irradiation plus protracted venous infusion (PVI) 5-FU radiosensitization vs PVI 5-FU prior to and following pelvic irradiation plus PVI 5-FU radiosensitization vs bolus 5-FU with leucovorin calcium and levamisole prior to and following pelvic irradiation. II. Describe relapse patterns and tolerance associated with these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to type of prior surgery (abdominoperineal resection vs anterior resection), nodal status (N0 vs N1 vs N2-3), depth of tumor invasion (T1-2 vs T3 vs T4a vs T4b), time from surgery to study entry (20-45 days vs 46-70 days), participating center, and performance status (0-1 vs 2). Patients are randomized to one of three treatment arms. Arm I: Patients receive fluorouracil (5-FU) IV on days 1-5 and 29-33. 5-FU is then given as a continuous infusion beginning on day 57 and continuing concurrently with radiotherapy for 5 weeks. Following a 28 day break from treatment patients receive 5-FU IV on days 1-5 of a 28 day course. Postradiotherapy treatment repeats for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive 5-FU IV continuously on days 1-42. 5-FU and radiotherapy are then administered as in arm II. Arm III: Patients receive leucovorin calcium (CF) IV followed by 5-FU IV on days 1-5 and 29-33. Patients also receive oral levamisole twice daily on days 1-3, 15-17, 29-31, and 43-45. CF IV and 5-FU IV are then given on days 57-60 and 85-88 concurrently with radiotherapy. Following a 28 day break from treatment patients receive CF IV and 5-FU IV on days 1-5 and 29-33 and oral levamisole twice daily on days 1-3, 15-17, 29-31, and 43-45 in the absence of disease progression or unacceptable toxicity. All patients receive radiotherapy 5 days per week for 5 weeks starting on day 57. Patients are followed every 4 months for 2 years, then every 6 months for 4 years, and then annually until death.

PROJECTED ACCRUAL: A total of 1,800 patients (600 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage II or III adenocarcinoma of the rectum Tumor extends through the bowel wall and into perirectal fat or soft tissue (TNM T3-4, N0, M0) Nodes are involved with tumor (TNM T1-4, N1-3, M0) Tumor completely resected en bloc with no gross or microscopic evidence of residual disease Circumferential (radial) margins of resected adherent tumors must be specifically documented free of disease (with the sole exception of extraperitoneal serosal margins) No evidence of metastasis No regional nodal metastases (metastases outside of the pelvis) that cannot be resected en bloc with the primary lesion No distant peritoneal metastases (metastases that are not a direct extension from the primary tumor) even if grossly resected (direct extension into another structure permitted) Abdominopelvic CT required unless: Bilirubin, SGOT, and alkaline phosphatase are within normal limits, AND Operative report describes liver as normal on exploration No tumors of colonic origin, i.e.: Lower edge of the tumor is below the peritoneal reflection or a portion of the tumor is retroperitoneally located (usually posteriorly) as defined by the surgeon at laparotomy OR Lower margin of the tumor is 12 cm or less from the anal verge by proctoscopic exam No prior history of rectal cancer No stage II or III cancers of the extrapelvic colon within the past 5 years Complete surgical resection at least 5 years prior to protocol registration allowed provided no other therapy was administered Synchronous modified stage I or IIa colorectal cancer (no nodal involvement or penetration through the muscularis propria) that has been completely resected allowed Registration between 20 and 70 days after the definitive surgical procedure required Chemotherapy must begin no later than day 70 following surgery Concurrent registration on protocol SWOG-9419 allowed for patients with adequate tissue samples

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: SWOG 0-2 Hematopoietic: WBC at least 4,000/mm3 Platelet count normal Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Alkaline phosphatase no greater than 2 times ULN Renal: Not specified Other: No chronic ulcerative colitis No other serious medical illness that would preclude protocol therapy No psychiatric condition that would preclude informed consent No noncolorectal malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Adequately treated carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics Other: No other concurrent antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1917 (Actual)
Dates: Start 1994-03; Primary Completion 2006-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Survival and Relapse-free survival | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Smalley, MD, Study Chair — University of Kansas; Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center; Jaffer A. Ajani, MD, Study Chair — M.D. Anderson Cancer Center; Michael J. O'Connell, MD, Study Chair — Mayo Clinic; Anthony LA Fields, MD, FRCPC, Study Chair — Cross Cancer Institute at University of Alberta; Robert J. Mayer, MD, FACP, Study Chair — Dana-Farber Cancer Institute
Locations (37):
- United States (35):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Ulrich CM, Rankin C, Holmes RS, et al.: Polymorphisms in folate-metabolizing enzymes and response to 5-fluorouracil among stage II or III rectal cancer patients (SWOG 9304). [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-309, 2008.
- [Result] Zhang W, Rankin CJ, Danenberg KD, et al.: An update of pharmacogenetic analysis of adjuvant rectal cancer patients treated with 5-fluorouracil and pelvic radiation in a phase III intergroup trial (INT-0144, SWOG 9304). [Abstract] J Clin Oncol 26 (Suppl 15): A-4115, 2008.
- [Result] Zhang W, Rankin C, Nagashima F, et al.: Pharmacogenetic analysis of stage II/III rectal cancer patients treated with 5-fluorouracil and pelvic radiation in a phase III intergroup trial (INT-0144, SWOG 9304). [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-300, 2008.
- [Result] Smalley SR, Benedetti JK, Williamson SK, Robertson JM, Estes NC, Maher T, Fisher B, Rich TA, Martenson JA, Kugler JW, Benson AB 3rd, Haller DG, Mayer RJ, Atkins JN, Cripps C, Pedersen J, Periman PO, Tanaka MS Jr, Leichman CG, Macdonald JS. Phase III trial of fluorouracil-based chemotherapy regimens plus radiotherapy in postoperative adjuvant rectal cancer: GI INT 0144. J Clin Oncol. 2006 Aug 1;24(22):3542-7. doi: 10.1200/JCO.2005.04.9544. PMID 16877719
- [Result] Smalley SR, Benedetti J, Williamson S, et al.: Intergroup 0144 - phase III trial of 5-FU based chemotherapy regimens plus radiotherapy (XRT) in postoperative adjuvant rectal cancer. Bolus 5-FU vs prolonged venous infusion (PVI) before and after XRT + PVI vs bolus 5-FU + leucovorin (LV) + levamisole (LEV) before and after XRT + bolus 5-FU + LV. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1006, 2003.